CLINICAL TRIAL: NCT00311428
Title: A Phase IV, Observer-Blind, Randomized, Parallel Groups, Single-Center, Exploratory Clinical Study to Evaluate the Immunogenicity and Safety of Two 0.25 mL Intramuscular Doses of Three Commercially Available Influenza Vaccines in Healthy Subjects Aged 6 to <36 Months.
Brief Title: Safety and Immunogenicity of Three Commercially Available Influenza Vaccines in Children Aged 6 to <36 Months
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M71P1; EUDRACT: 2004-001952-35
Record Dates: First submitted 2006-04-03; First posted 2006-04-06 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Influenza
Keywords: Influenza; Children; Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza

SUMMARY:
This phase IV protocol is designed to evaluate the safety, clinical tolerability and immunogenicity of the 2005-2006 formulation of three widely used conventional influenza vaccines in children aged 6 to 35 months

ELIGIBILITY:
Inclusion Criteria:

* children of 6 months to <36 months of age, whose parents or legal guardians have given written informed consent prior to study entry

Exclusion Criteria:

* Any severe acute respiratory disease and infections requiring systemic antibiotic or antiviral therapy ongoing or resolved within 30 days prior to study start (chronic antibiotic therapy for urinary tract prophylaxis is acceptable)
* Other serious diseases such as: cancer, autoimmune disease (including rheumatoid arthritis), diabetes mellitus, chronic pulmonary disease, acute or progressive hepatic or renal disease, surgery planned during the study period.
* Known or suspected impairment/alteration of immune function
* History of hypersensitivity to any component of the study vaccine, egg products or other vaccine component, or impairment/alteration of immune function

Ages: 6 Months to 35 Months | Sex: All
Age Groups: Child
Enrollment: 270
Dates: Start 2005-10

PRIMARY OUTCOMES:
Seroprotection, GMR's and Seroconversion rate at day 0 and day 50 following vaccination.

SECONDARY OUTCOMES:
Solicited Local and Systemic Reactions Within 6 Days Following Each Vaccination And Adverse Events Thought the Study.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines Information Services, Study Chair — Novartis Vaccines & Diagnostics
Locations (1):
- University of Tampere Medical School, Tampere, Finland